CLINICAL TRIAL: NCT06401486
Title: Video Versus Direct Laryngoscopy for Double-lumen Tube Tracheal Intubation in Thoracic Surgery
Brief Title: DOuble-Lumen Intubation With VIdeolaryngoscopy
Acronym: DoLVi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Proffesor, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DoLVi trial
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Intubation Complication; Intubation; Difficult or Failed; Anesthesia; Videolaryngoscopy
Keywords: videolaryngoscopy; tracheal intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Videolaryngoscope group (Active Comparator): For patients assigned to the videolaryngoscope Group, the operator will use a videolaryngoscope on the first laryngoscopy attempt.
  Interventions: Device: Videolaryngoscope
- Macintosh laryngoscope Group (Active Comparator): For patients assigned to the laryngoscope Group, the operator will use a Macintosh laryngoscope on the first laryngoscopy attempt.
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: Videolaryngoscope — For patients assigned to the videolaryngoscope Group, the operator will use a video laryngoscope on the first laryngoscopy attempt.
  Arms: Videolaryngoscope group
Device: Macintosh laryngoscope — For patients assigned to the laryngoscope Group, the operator will use a Macintosh laryngoscope on the first laryngoscopy attempt.
  Arms: Macintosh laryngoscope Group

SUMMARY:
Tracheal intubation (TI) is one of the fundamental and most recognized techniques in Anesthesiology, also essential in all units treating urgent pathology and critical patients. It involves advancing a tube through the vocal cords into the trachea to ventilate the patient. In thoracic surgery, it is often necessary to achieve lung isolation, ventilating only one lung while the operated lung remains collapsed and immobile. To achieve this, it is common to intubate the patient with a special tube: a double-lumen tube (DLT), larger than usual because it provides two ventilation channels, one for each lung.

Tracheal intubation with a DLT presents some peculiarities: its larger size and stiffness make manipulation and orientation in the oropharynx difficult. It has a curve at its distal end (the bronchial lumen) designed to slide into the left or right main bronchus as needed. The fact that the DLT passes between the vocal cords does not ensure its proper placement and function. Therefore, DLT intubation requires practice and experience, both to slide it between the vocal cords and to position it properly.

The classic technique for DLT intubation is "Direct Laryngoscopy" (DL). A traditional laryngoscope with a Macintosh blade is used to move the upper airway structures aside to allow direct visualization of the glottis. In recent years, to facilitate tracheal intubation, different videolaryngoscopes have appeared. A videolaryngoscope is a device similar to a traditional laryngoscope that allows, thanks to an image sensor located at its end, indirect visualization of the glottis on an integrated or external screen.

There is strong evidence for the benefit of using a VL over traditional DL in single-tube intubation in adult patients. However, although the use of VL for DLT intubation is becoming more common, there are few studies with small sample sizes comparing VL to DL for DLT intubation, so the evidence of its advantages or disadvantages is of low quality. It could improve glottic exposure and the percentage of success on the first attempt, although there is a possibility of increased tube malposition incidence and delayed intubation.

Therefore, Investigators propose a prospective, multicenter, randomized study comparing the traditional Macintosh blade laryngoscope (direct laryngoscopy) with the videolaryngoscope to facilitate orotracheal intubation with double-lumen tube in patients scheduled for thoracic surgery requiring lung isolation.

DETAILED DESCRIPTION:
The purpose of this prospective multicenter randomized study is to compare successful intubation on the first attempt with the Macintosh laryngoscope vs the videolaryngoscope for double-lumen tube tracheal intubation in thoracic surgery. Investigators hypothesize that tracheal intubation using the videolaryngoscope will improve the frequency of successful intubation on the first attempt.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients admitted to any of the participating hospitals in the study who are undergoing thoracic surgery.
* Need for intubation with a double-lumen tube.

Exclusion Criteria:

* Pregnant or lactating women.
* Individuals who do not have the capacity to understand their participation in the study.
* Need for tracheal intubation with a device other than videolaryngoscopy or direct laryngoscopy (fiberoptic bronchoscope, tracheostomy...).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 916 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Number of intubations with successful intubation on the first attempt | Duration of procedure (minutes)
  The primary outcome is defined as placement of a double lumen tube in the trachea with a single insertion of a videolaryngoscope blade into the mouth and either a single insertion of a double lumen tube into the mouth.

SECONDARY OUTCOMES:
Successful intubation | Duration of procedure (minutes)
  Successful placement of a double lumen tube in the trachea
Incidence of "easy intubation" | Duration of procedure (minutes)
  Easy intubation is defined as a patient with Cormack-Lehane I-II glottic view and intubation on the first attempt.

OTHER OUTCOMES:
Number of laryngoscopy attempts | Duration of procedure (minutes)
  Number of laryngoscopy attempts
Number of attempts to cannulate the trachea with an endotracheal tube | Duration of procedure (minutes)
  Number of attempts to cannulate the trachea with an endotracheal tube
Duration of laryngoscopy and tracheal intubation | Duration of procedure (minutes)
  The interval (in seconds) between the first insertion of a laryngoscope blade into the mouth and the final placement of a double lumen tube in the trachea.
Reason for failure to intubate on the first attempt | Duration of procedure (minutes)
  Reason for failure among those who did not meet the primary outcome (successful intubation on the first attempt):
  * Inadequate view of the larynx
  * Inability to intubate the trachea with an endotracheal tube
  * Inability to cannulate the trachea with a bougie
  * Attempt aborted due to change in patient condition (e.g., worsening hypoxemia, hypotension, bradycardia, vomiting, bleeding)
  * Technical failure of the laryngoscope (e.g., battery, light source, camera, screen)
  * Other
Operator-assessed difficulty of intubation | Duration of procedure (minutes)
  Operator-assessed difficulty of intubation
  * without difficulty
  * mild difficulty
  * moderate difficulty
  * severe difficulty
Modified Cormack-Lehane grade of glottic view | Duration of procedure (minutes)
  Modified Cormack-Lehane grade of glottic view:
  * I: full view of the glottis
  * IIa: partial view of the glottis
  * IIb: arytenoid or posterior part of the vocal cords just visible
  * III: only epiglottis visible
  * IV: neither glottis nor epiglottis visible Cormack-Lehane grade of glottic view
Need for additional airway equipment | Duration of procedure (minutes)
  Airway equipment: bougie, stylet, other videolaryngoscope, others.
Need to change the device for intubation | Duration of procedure (minutes)
  Need to replace by another videolaryngoscope, a different angled blade, requirement for a fiberoptic bronchoscope...).
Use of external laryngeal pressure | Duration of procedure (minutes)
  External laryngeal pressure
Malposition of the double lumen endotracheal tube | Duration of procedure (minutes)
  Malposition of the double lumen endotracheal tube
Incidence of Dysphonia, hoarseness, or sore throat in the first 24 hours. | 24 hours after intubation
  Incidence of Dysphonia, hoarseness, or sore throat in the first 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada, Ph.D., Principal Investigator — Clinical University Hospital of Santiago de Compostela
Locations (4):
- Spain (4):
  - Complexo Hospitalario Universitario de A Coruña, A Coruña
  - Complexo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario La Fe de Valencia, Valencia
  - Complexo Hospitalario Universitario Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karczewska K, Bialka S, Smereka J, Cyran M, Nowak-Starz G, Chmielewski J, Pruc M, Wieczorek P, Peacock FW, Ladny JR, Szarpak L. Efficacy and Safety of Video-Laryngoscopy versus Direct Laryngoscopy for Double-Lumen Endotracheal Intubation: A Systematic Review and Meta-Analysis. J Clin Med. 2021 Nov 25;10(23):5524. doi: 10.3390/jcm10235524. PMID 34884226
- [Background] Kim YS, Song J, Lim BG, Lee IO, Won YJ. Different classes of videoscopes and direct laryngoscopes for double-lumen tube intubation in thoracic surgery: A systematic review and network meta-analysis. PLoS One. 2020 Aug 28;15(8):e0238060. doi: 10.1371/journal.pone.0238060. eCollection 2020. PMID 32857788
- [Background] Liu TT, Li L, Wan L, Zhang CH, Yao WL. Videolaryngoscopy vs. Macintosh laryngoscopy for double-lumen tube intubation in thoracic surgery: a systematic review and meta-analysis. Anaesthesia. 2018 Aug;73(8):997-1007. doi: 10.1111/anae.14226. Epub 2018 Feb 6. PMID 29405258